CLINICAL TRIAL: NCT01512550
Title: Evaluation of the Importance in Restoring Biomechanical Correct Hip Anatomy During THA. A Prospective, Randomized and Controlled Study Evaluated by RSA, CT and Gait Analysis
Brief Title: Importance of Restoring Biomechanical Correct Hip Anatomy During Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Gunnar Flivik, Associate Professor, MD PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HipBiomech-SK
Record Dates: First submitted 2012-01-06; First posted 2012-01-19 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis
Keywords: Radiostereometric Analysis (RSA); Total hip arthroplasty (THA); Hip anatomy; Hip biomechanics
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- instrumented hip guide technique (Active Comparator): A mechanical device used to measure and decide how the hip prosthesis (ABG II modular) should be implanted
  Interventions: Procedure: GF hip guide; Device: ABG II modular femoral component
- conventional measuring technique (No Intervention): Standard way of implanting the prosthesis (ABG II standard) without special measuring device or computer navigation technique
- computer assisted navigation (Active Comparator): A method to use computer navigation when positioning and sizing the hip prosthesis (ABG II modular).
  Interventions: Procedure: Stryker Navigation System; Device: ABG II modular femoral component

INTERVENTIONS:
Procedure: GF hip guide — Using GF hip guide to measure and control the peroperative positioning of the hip stem
  Other Names: Instrument designed by the investigators
  Arms: instrumented hip guide technique
Procedure: Stryker Navigation System — Using Orthomap Modular Hip Software to navigate the operation
  Other Names: Stryker Orthomap Hip Navigation System
  Arms: computer assisted navigation
Device: ABG II modular femoral component — A hip prosthesis made by Stryker. It has the same basic shape as the ABG II femoral component but has a modular neck system allowing it to better follow the patient specific hip anatomy regarding offset, varus-valgus angle and rotation in the anteroposterior plane.
  Other Names: ABG™II modular Cementless Hip System
  Arms: computer assisted navigation; instrumented hip guide technique

SUMMARY:
The purpose of this prospective, randomized study is to evaluate the importance of restoring the exact individual hip biomechanics during total hip arthroplasty.

DETAILED DESCRIPTION:
This prospective, controlled and randomized study aims at evaluating the correlation between postoperative hip prosthesis migration and the achieved exactness of biomechanical restoration of hip mechanics during total hip arthroplasty (THA). The main objective is to find out how close the result from the surgery can come to a preferred prosthesis position and whether this makes any difference in terms of loosening, functionality and quality of life for the patient. The prosthesis positioning is performed with either (1) computer assisted navigation, (2) instrumented hip guide measuring devise alignment technique or (3) conventional non-instrumented measuring technique. The ABG II stem system (Stryker) will be used in the modular version for group 1 and 2 and the non-modular version in group 3. Before each operation the investigators will perform exact measurements of anatomical variables using preoperative radiographs (maximum 8 weeks old) and computed tomography images (CT)(taken 3-4 weeks preoperatively). While applying these measurements the investigators will try to preserve the patient´s individual biomechanical situation, most often as compared to the healthy contralateral hip. The variables to be analysed are anteversion of the femoral neck, offset and leg length. This preoperative hip analysis combined with the use of a templating system will give the data needed for component choice and exact positioning of the ABG II hip prosthesis. 75 patients will be randomized into the three groups (25+25+25). The patients will be followed with RadioStereometric Analysis (RSA) for two years (directly postoperatively, 14 days, 3 months, 1 year and 2 years). There will be a second CT scan 1 year postoperatively to measure the actual achieved position. In completion hip specific and general health questionnaires will be used to evaluate patient satisfaction and outcome. All patients will be subject to 3-Dimensional (3-D) gait analysis 3-4 weeks prior to surgery and after one year. The results of the gait analysis will be correlated to the achieved restoration of the hip anatomy and biomechanics. The investigators aim is to improve the fundamental understanding of the hip biomechanics in patients undergoing THA. Will physical performance improve when the individual hip biomechanics is better restored, and in which way and to what extent?

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis (OA) of the hip necessitating primary total hip arthroplasty (THA)
* Male and non-pregnant female patients
* Hip bone quality and morphology suitable for uncemented THA
* Age up to 75 years old at the inclusion time of the study
* Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up.
* Patients who are capable of, and have given informed consent for participation in the study.

Exclusion Criteria:

* Rheumatoid arthritis
* Malignant disease
* Severe osteoporosis
* Patients with active infection
* Patients with malignancy
* Prior major surgery in the hip to be operated on
* Peroperative fracture
* Hip prosthesis or grossly distorted hip anatomy in the contralateral hip.
* Ongoing corticosteroid (oral) or immunosuppressive medication
* Personal disorders (dementia, alcohol or drug abuse etc) suspected of making completion of the trial uncertain.
* Patients with concurrent illnesses which are likely to affect their outcome.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Radiostereometric Analysis (RSA) | First postoperative day(reference examination), 14 days, 3 months, 1 and 2 years
  This will measure the change in migration (translation and rotation around the x-, y- and z-axis of the hip) over time from baseline which is the direct postoperative examination and up to 2 years postoperatively. The migration pattern over a 2-year period can predict the long-term fate of the prosthesis

SECONDARY OUTCOMES:
Gait analysis | Preoperatively (3-4 weeks) and 1 year postoperatively
  This will measure how the patients gait pattern has changed from preoperatively when the patient had symptoms from osteoarthritis and 1 year postoperatively when everything has healed and the new hip prosthesis should have full effect on function and pain relive.
Computer Tomography (CT) | Preoperatively (3-4 weeks) and 1 year postoperatively
  This will measure how much the anatomy has changed from preoperatively to after the new hip prosthesis has been put in. Are the goals of hip anatomy restoration achieved? The main measurements will be leg length, global offset and rotation of femoral neck.
General and hip specific health questionnaires | preoperatively (3-4 weeks), 1 and 2 years postoperatively
  Hip disability and Osteoarthritis Outcome Score (HOOS) - this is a hip specific questionnaire that will measure how the operation has affected the patients function and pain situation over time.
  EuroQol (EQ-5D) - a standardized instrument for use as measure of general health outcome over time

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Flivik, MD PhD, Principal Investigator — Dept of Orthopedics, Skane University Hospital, Lund University, Sweden
Locations (1):
- Department of Orthopedics, Skane University Hospital, Lund University, Lund, Sweden

REFERENCES:
- [Derived] Esbjornsson AC, Kiernan S, Mattsson L, Flivik G. Geometrical restoration during total hip arthroplasty is related to change in gait pattern - a study based on computed tomography and three-dimensional gait analysis. BMC Musculoskelet Disord. 2021 Apr 20;22(1):369. doi: 10.1186/s12891-021-04226-4. PMID 33879123
- [Derived] Kiernan S, Kaptein B, Flivik C, Sundberg M, Flivik G. Unexpected varus deformity and concomitant metal ion release and MRI findings of modular-neck hip stems: descriptive RSA study in 75 hips with 8 years' follow-up. Acta Orthop. 2021 Feb;92(1):67-73. doi: 10.1080/17453674.2020.1853387. Epub 2020 Dec 10. PMID 33297800
- [Derived] Kiernan S, Geijer M, Sundberg M, Flivik G. Effect of symmetrical restoration for the migration of uncemented total hip arthroplasty: a randomized RSA study with 75 patients and 5-year follow-up. J Orthop Surg Res. 2020 Jun 17;15(1):225. doi: 10.1186/s13018-020-01736-0. PMID 32552711